CLINICAL TRIAL: NCT02244788
Title: Humanitarian Use of AVANTA Orthopaedics Proximal Interphalangeal Joint
Status: Available | Type: Expanded Access
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-059
Record Dates: First submitted 2014-09-16; First posted 2014-09-19 (Estimated); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Arthroplasty of the PIP Joint

INTERVENTIONS:
Device: SR™ PIP — SR™ PIP

SUMMARY:
The purpose of this study is to allow patients to undergo surgery with the SR™ PIP (Proximal Interphalangeal) Implants for finger arthritis. This is NOT a research study, but rather, a requirement by the FDA for humanitarian use of device

DETAILED DESCRIPTION:
The purpose of this IRB approved study is to allow patients to undergo surgery with the SR™ PIP (Proximal Interphalangeal) Implants. This is NOT a research study, but rather, a requirement by the FDA for humanitarian use of device. Use of the SR™ PIP is approved for humanitarian use by the FDA when either the patient is in need of a revision of failed PIP prothesis(es) or the patient expects to place his/her hand under loading situation which preclude the use of an alternative implant in the painful osteo-arthritic and post traumatic arthritic PIP joint.

ELIGIBILITY:
Inclusion Criteria:

* patient is in need of a revision of failed PIP prosthesis(es)
* patient expects to place his/her hands under loading situations which preclude the use of an alternative implant in the painful osteo-arthritic and post traumatic arthritic PIP joint

Exclusion Criteria:

* patient is not in need of a revision of a failed PIP prothesis(es)
* patient is eligible to use an alternative implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Edward Athanasian, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States